CLINICAL TRIAL: NCT04179006
Title: Effects of Nutrients Supplementation in Antidepressant Treated Depressive Disorder Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Cheng-Kung University Hospital (Other)
Collaborators: Grape King Bio Ltd. (Industry)
Responsible Party: Principal Investigator, Po-See, Chen, Principal Investigator, Professor, Visiting Staff Psychiatrist of Department of Psychiatry, Professor (joint appointment) of Institute of Behavioral Medicine, National Cheng-Kung University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: B-BR-108-032
Record Dates: First submitted 2019-11-19; First posted 2019-11-26 (Actual); Last update posted 2021-09-10 (Actual); Status verified 2021-09

CONDITIONS: Depressive Disorder, Major
Keywords: Major depressive disorder; Supplement nutrients; Antidepressants
MeSH Terms: conditions — Depressive Disorder, Major

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- LF chocolate + antidepressant(s) (Active Comparator): Participants with LF chocolate add-on to their antidepressants regimen.
  Interventions: Dietary Supplement: LF/Erinacine A-enriched Hericium/Plain chocolate + antidepressant(s)
- Erinacine A-enriched Hericium chocolate + antidepressant(s) (Active Comparator): Participants with Erinacine A-enriched Hericium chocolate add-on to their antidepressants regimen.
  Interventions: Dietary Supplement: LF/Erinacine A-enriched Hericium/Plain chocolate + antidepressant(s)
- Plain chocolate + antidepressant(s) (Placebo Comparator): Participants with plain chocolate add-on to their antidepressants regimen.
  Interventions: Dietary Supplement: LF/Erinacine A-enriched Hericium/Plain chocolate + antidepressant(s)

INTERVENTIONS:
Dietary Supplement: LF/Erinacine A-enriched Hericium/Plain chocolate + antidepressant(s) — 3 pieces per day

SUMMARY:
This is a randomized, double-blind, placebo-controlled to evaluate the potential role of nutrients supplementation (LF chocolate /Erinacine A-enriched Hericium Erinaceus chocolate) on the therapeutic efficacy of antidepressants in major depressive disorder(MDD).

120 subjects who meet all the inclusion and exclusion criteria will be randomized into three categories, receiving 3 pieces of supplement nutrients-added or plain chocolates per day for a period of 24 weeks in total. The three categories are as follow:

1. LF chocolate
2. Erinacine A-enriched Hericium Erinaceus chocolate
3. Plain chocolate without any supplementary nutrients added (placebo group) These MDD patients will continue their antidepressant regimen throughout the study.

Symptom rating, blood samples for antidepressant-related/depressive disorder-related genome profiles identification, as well as for biomarkers assessment for metabolic indices, questionnaires and tests for psychosocial variables identification and patient's cognitive and social cognitive function or performance determination, will be carried out before and at certain time points within the 24-week tracking period. Patient's fecal samples will be acquired to recognize and to distinguish the alterations of these MDD patients microbiota profiles over the 24-week period.

DETAILED DESCRIPTION:
Major depressive disorder (MDD) is a common, severe, and often life-threatening illness that involves the body, mood, and thoughts. Recent reports suggested that immune dysfunction could be linked with cognitive impairment and metabolic comorbidities, and accumulating evidence suggested that the regulation of the microbiota- gut-brain axis has been shown to impact inflammation and to affect brain function.

This randomized, double-blind, placebo-controlled is to evaluate the potential role of nutrients supplementation (LF chocolate /Erinacine A-enriched Hericium Erinaceus chocolate) on the therapeutic efficacy of antidepressants in major depressive disorder(MDD). 120 MDD outpatients (aged 20-70 years) from the National Cheng Kung University Hospital who meet the Diagnostic and Statistical Manual of mental disorders, Fifth Edition (DSM-5) and Hamilton Rating Scale for Depression (HAMD) scores ≥ 7, receiving fluoxetine or venlafaxine so as SSRI or SNRI antidepressants will be enrolled.

Subjects who meet all the inclusion and exclusion criteria will be randomized into three categories, with 40 subjects each, receiving 3 pieces of supplement nutrients-added or plain chocolates (placebo) manufactured by GRAPE KING BIO LTD per day for a period of 24 weeks in total. The three categories are as follow:

1. LF chocolate
2. Erinacine A-enriched Hericium Erinaceus chocolate
3. Plain chocolate without any supplementary nutrients added (placebo group) These MDD patients will continue their antidepressant regimen throughout the study. Follow-up visits will be arranged at week no. 0, 2, 4, 8, 12, 16, 20 and 24, in which week no. 0, 4, 12 and 24 will be the four most important re-visit timing.

Various assessments or tests will be arranged in these 24-week period. Symptom rating with 17-item Hamilton Rating Scale for Depression (HAM-D) by psychiatrist will be done at every visits. Blood samples for antidepressant-related/depressive disorder-related genome profiles identification, as well as for biomarkers assessment for metabolic indices, will be obtained at week no. 0, 4, 12 and 24. Questionnaires aimed for psychosocial variables (environmental factors) identification including social support scales (SSS), quality of life scale (QOLs) and Recent life changes questionnaire (RCLQ) will be self-answered by patients. Continuous Performance Test (CPT), finger-Tapping Test (FPT) and Wisconsin Card Sorting Test (WCST) will be utilized to evaluate their cognitive performance. Mayer-Salovey-Caruso emotional Intelligent Test (MSCEIT) will help in social cognitive function assessment. Patient's fecal samples will be acquired at week no. 0, 4, 12 and 24 to recognize and to distinguish the alterations in MDD patients microbiota profiles.

ELIGIBILITY:
Inclusion Criteria:

* Major depressive disorder (MDD) outpatients meet DSM- criteria
* Hamilton Rating Scale for Depression (HAM-D) ≥ 7
* Start to receive fluoxetine or venlafaxine or those who have received the SSRI or SNRI antidepressants

Exclusion Criteria:

* (A) had DSM-5 diagnosis for substance abuse within the past three months;
* (B) had taken monoamine oxidase inhibitors;
* (C) had an organic mental disorder, mental retardation, dementia, or other diagnosed neurological illness;
* (D) had a surgical condition or a major physical illness;
* (E) pregnant or breast-feeding.

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2019-11-14 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in participant's Hamilton Rating Scale for Depression (HAM-D) score | week no. 0, 2, 4, 8, 12, 16, 20, 24
  Depressive symptom rating; 21 items int total, eight items are scored on a 5-point scale, ranging from 0 = not present to 4 = severe, while nine are scored from 0-2; [higher scores denote worse symptoms/signs of depression]
Change in participant's BW(kg), Height(cm), Waist circumference(cm), BMI (kg/m2) | week no. 0, 2, 4, 8, 12, 16, 20, 24
  Metabolic indices; BW (to the nearest 0.1 kg), height (to the nearest 0.1 cm), and waist circumference (to the nearest 0.1 cm), weight and height will be combined to report BMI in kg/m^2
Change in participant's Glucose profiles | week no. 0, 4, 12, 24
  Metabolic indices; HbA1c(%)+Fasting plasma glucose (mg/dl)+Fasting serum insulin concentrations (uIU/ml)+Homeostasis model assessment-estimated insulin resistance (HOMA-IR) index+Homeostasis model of assessment for pancreatic β-cell secretory function (HOMA-β) {HOMA- IR= [fasting plasma insulin level (uIn/ml)*fasting plasma glucose level (mg/dl)/405]; HOMA- IR ≥2.5 => Insulin resistance (+)} {HOMA-β= (360× fasting serum insulin [uIn/ml]) / (fasting plasma glucose [mg/dL] -63)}
Change in participant's Fasting serum leptin level (ng/mL) | week no. 0, 4, 12, 24
  Metabolic indices
Change in participant's Fasting serum lipid profiles | week no. 0, 4, 12, 24
  Metabolic indices; including Fasting total cholesterol(mg/dL), High density lipoprotein (HDL) cholesterol(mg/dL), Low-density lipoprotein (LDL) cholesterol(mg/dL), Triglyceride (TG) concentration(mg/dL)
Change in participant's Cortisol(ug/dL) level | week no. 0, 4, 12, 24
  Metabolic indices
Change in participant's C-peptide(ng/dL) | week no. 0, 4, 12, 24
  Metabolic indices
Change in participant's Inflammatory cytokines levels | week no. 0, 4, 12, 24
  Metabolic indices; Fasting plasma C-reactive protein (CRP) level (pg/mL) + Oxytocin(pg/mL) + Leptin(mg/mL)
Change in participants's Quality of life scale (QOLs) scores [WHOQOL-BREF] | week no. 0, 4, 12, 24
  Psychosocial variables as environment factors; Quality of Life Scale developed through the World Health Organization (WHOQOL-BREF) & Health-Related Quality of Life (HRQOL) questionnaires will be used as assessment tools WHOQOL-BREF: 4 domains will be assessed, consists of 1. Physical Health 2. Psychological 3. Social Relationship 4. Environment; [higher scores in each domains denote higher quality of life]
Change in participants's Quality of life scale (QOLs) scores [HRQOL] | week no. 0, 4, 12, 24
  Psychosocial variables as environment factors; Quality of Life Scale developed through the World Health Organization (WHOQOL-BREF) & Health-Related Quality of Life (HRQOL) questionnaires will be used as assessment tools HRQOL: 4 domains will be assessed, consists of 1. Physical Health 2. Psychological 3. Level of independence 4. Social Relationship [higher scores in each domains denote higher quality of life]
Change in participant's Cognitive performance | week no. 0, 12, 24
  Continuous Performance Test (CPT)[visual information processing & attentive capacity], Finger Tapping Test (FPT), Wisconsin Card-Sorting Test (WCST)
Change in participant's Social cognitive functional performance | week no. 0, 12, 24
  Mayer-Salovey-Caruso emotional Intelligence Test (MSCEIT) scores; perceiving + facilitating + understanding + managing emotion
Change in participant's Microbiota profiles | week no. 0, 12, 24
  Fecal samples; Types of microorganisms + no. of colonies (colony-forming unit, CFU)

CONTACTS AND LOCATIONS:
Locations (1):
- National Cheng-Kung University, Tainan, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Byers AL, Yaffe K. Depression and risk of developing dementia. Nat Rev Neurol. 2011 May 3;7(6):323-31. doi: 10.1038/nrneurol.2011.60. PMID 21537355
- [Background] Gorska-Ciebiada M, Saryusz-Wolska M, Ciebiada M, Loba J. Mild cognitive impairment and depressive symptoms in elderly patients with diabetes: prevalence, risk factors, and comorbidity. J Diabetes Res. 2014;2014:179648. doi: 10.1155/2014/179648. Epub 2014 Nov 9. PMID 25431771
- [Background] Chang HH, Chi MH, Lee IH, Tsai HC, Gean PW, Yang YK, Lu RB, Chen PS. The change of insulin levels after six weeks antidepressant use in drug-naive major depressive patients. J Affect Disord. 2013 Sep 5;150(2):295-9. doi: 10.1016/j.jad.2013.04.008. Epub 2013 May 9. PMID 23664565
- [Background] Howren MB, Lamkin DM, Suls J. Associations of depression with C-reactive protein, IL-1, and IL-6: a meta-analysis. Psychosom Med. 2009 Feb;71(2):171-86. doi: 10.1097/PSY.0b013e3181907c1b. Epub 2009 Feb 2. PMID 19188531
- [Background] Chang HH, Lee IH, Gean PW, Lee SY, Chi MH, Yang YK, Lu RB, Chen PS. Treatment response and cognitive impairment in major depression: association with C-reactive protein. Brain Behav Immun. 2012 Jan;26(1):90-5. doi: 10.1016/j.bbi.2011.07.239. Epub 2011 Aug 4. PMID 21839826
- [Background] Hiles SA, Baker AL, de Malmanche T, Attia J. Interleukin-6, C-reactive protein and interleukin-10 after antidepressant treatment in people with depression: a meta-analysis. Psychol Med. 2012 Oct;42(10):2015-26. doi: 10.1017/S0033291712000128. Epub 2012 Feb 16. PMID 22336436
- [Background] Fabbri C, Porcelli S, Serretti A. From pharmacogenetics to pharmacogenomics: the way toward the personalization of antidepressant treatment. Can J Psychiatry. 2014 Feb;59(2):62-75. doi: 10.1177/070674371405900202. PMID 24881125
- [Background] Antypa N, Drago A, Serretti A. Genomewide interaction and enrichment analysis on antidepressant response. Psychol Med. 2014 Mar;44(4):753-65. doi: 10.1017/S0033291713001554. Epub 2013 Jul 1. PMID 23809733
- [Background] Biernacka JM, Sangkuhl K, Jenkins G, Whaley RM, Barman P, Batzler A, Altman RB, Arolt V, Brockmoller J, Chen CH, Domschke K, Hall-Flavin DK, Hong CJ, Illi A, Ji Y, Kampman O, Kinoshita T, Leinonen E, Liou YJ, Mushiroda T, Nonen S, Skime MK, Wang L, Baune BT, Kato M, Liu YL, Praphanphoj V, Stingl JC, Tsai SJ, Kubo M, Klein TE, Weinshilboum R. The International SSRI Pharmacogenomics Consortium (ISPC): a genome-wide association study of antidepressant treatment response. Transl Psychiatry. 2015 Apr 21;5(4):e553. doi: 10.1038/tp.2015.47. PMID 25897834
- [Background] Rogers GB, Keating DJ, Young RL, Wong ML, Licinio J, Wesselingh S. From gut dysbiosis to altered brain function and mental illness: mechanisms and pathways. Mol Psychiatry. 2016 Jun;21(6):738-48. doi: 10.1038/mp.2016.50. Epub 2016 Apr 19. PMID 27090305
- [Background] Soto M, Herzog C, Pacheco JA, Fujisaka S, Bullock K, Clish CB, Kahn CR. Gut microbiota modulate neurobehavior through changes in brain insulin sensitivity and metabolism. Mol Psychiatry. 2018 Dec;23(12):2287-2301. doi: 10.1038/s41380-018-0086-5. Epub 2018 Jun 18. PMID 29910467
- [Background] Jiang H, Ling Z, Zhang Y, Mao H, Ma Z, Yin Y, Wang W, Tang W, Tan Z, Shi J, Li L, Ruan B. Altered fecal microbiota composition in patients with major depressive disorder. Brain Behav Immun. 2015 Aug;48:186-94. doi: 10.1016/j.bbi.2015.03.016. Epub 2015 Apr 13. PMID 25882912